CLINICAL TRIAL: NCT04375085
Title: A Non-Randomized, Post Marketing Clinical Follow-Up (PMCF) Study of the DESyne X2 Novolimus Eluting Coronary Stent System in the Treatment of Patients With de Novo Native Coronary Artery Lesions
Brief Title: DESyne X2 Post Market Follow-up Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment was delayed and could not be completed as planned
Sponsor: Elixir Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELX-CL-1705
Record Dates: First submitted 2020-04-29; First posted 2020-05-05 (Actual); Results first posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Disease
Keywords: coronary stent; percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- DESyne X2 Novolimus Eluting Coronary Stent System (Other)
  Interventions: Device: Percutaneous Coronary Intervention

INTERVENTIONS:
Device: Percutaneous Coronary Intervention — Percutaneous Coronary Intervention

SUMMARY:
A single-arm post-market clinical follow-up study to confirm that the DESyne X2 delivery system performs similarly to the DESyne delivery system.

DETAILED DESCRIPTION:
A single-arm post-market follow up study (PMCF) comparing the DESyne X2 PMCF data to the historic DESyne acute performance data to confirm the performance of the DESyne X2 Novolimus Eluting Coronary Stent System with regards to the residual risks of lesion access and acute device implantation through visually-assessed angiographic endpoints and physician feedback.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be ≥ 18 years of age.
2. The patient must have stable angina pectoris as defined by the Canadian Cardiovascular Society Classification, documented silent ischemia, acute coronary syndrome, or a positive functional study requiring treatment
3. The patient is considered a candidate for coronary stent implantation and has a planned intervention of up to two lesions located in separate major epicardial territories. Each lesion/vessel must meet the following criteria:

   1. De novo lesion
   2. The target lesion reference site must be visually estimated to be ≥ 2.5 mm and ≤ 4.0 mm in diameter
   3. The target vessel must be a major coronary artery or major branch with a visually estimated stenosis of ≥ 50% and < 100%.
   4. The visually estimated target lesion length must be ≤ 34 mm
   5. ≥ TIMI 1 coronary flow

Exclusion Criteria:

1. The patient has a known hypersensitivity or contraindication to aspirin, heparin, ticlopidine, clopidogrel, prasugrel or ticagrelor, heparin/bivalirudin, mTOR inhibitor class drugs, cobalt chromium alloy, methacrylate or polylactide polymer, or sensitivity to contrast which cannot be adequately premedicated
2. Women of childbearing potential who have not undergone surgical sterilization or are not post-menopausal (defined as amenorrheic for at least one year) as well as women who are pregnant or nursing
3. Previous placement of a stent within 10 mm distal to the target lesion
4. Previous placement of a stent proximal to the target lesion
5. Total occlusion or < TIMI 1 coronary flow in the target vessel
6. The proximal target vessel or target lesion is severely calcified by visual assessment
7. Aorto-ostial location, unprotected left main lesion location, or a lesion within 5 mm of the origin of the left anterior descending or left circumflex
8. Lesion involvement of a significant side branch (branch diameter > 2 mm) that would be covered by stenting
9. High probability that treatment other than PTCA or stenting will be required for treatment of the same lesion
10. The target lesion, or the target vessel proximal to the target lesion, contains thrombus
11. The patient has suffered a myocardial infarction within the past 72 hours and the CK or CK-MB has not returned to normal at the time of the index procedure
12. The patient is a recipient of a heart transplant
13. The patient has extensive peripheral vascular disease that precludes safe sheath insertion or extreme anti-coagulation
14. The patient is currently participating in another investigational device or drug study that has not completed the primary follow-up phase
15. Patients who are unable or unwilling to cooperate with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Kwong Wah Hospital, Hong Kong, Kowloon
  - Queen Elizabeth Hospital, Hong Kong, Kowloon
  - Tseung Kwan O Hospital, Hong Kong

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 49 Patients were enrolled at 3 investigational sites in Hong Kong between 1 Sep 2020 to 28 Dec 2021. The enrollment was halted at 49 of 100 patients due to slow enrollment.
Groups:
- DESyne X2 Novolimus Eluting Coronary Stent System: Enrollment of up to 100 patients with up to three de novo native coronary artery lesions receiving the DESyne X2 Novolimus Eluting Coronary Stent System (CSS).
Period: Overall Study
Arm/Group | DESyne X2 Novolimus Eluting Coronary Stent System
Started | 49
Completed | 49
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- DESyne X2 Novolimus Eluting Coronary Stent System: Enrollment of up to 100 patients with up to three de novo native coronary artery lesions measuring between 2.25 and 4.0 mm in diameter and less than or equal to 34 mm in length receiving the DESyne X2 Novolimus Eluting Coronary Stent System (CSS).
Arm/Group | DESyne X2 Novolimus Eluting Coronary Stent System
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 39
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Hong Kong | 49

OUTCOME MEASURES:

1. Primary Outcome: Acute Success
Description: attainment of final result with < 50% residual stenosis of the target site, using a DESyne X2 stent and standard pre-dilation catheters and post-dilatation catheters (if applicable)
Time Frame: during procedure
Measure: Count of Participants; unit: Participants
Groups:
- Acute Success: The DESyne X2 Novolimus Eluting Coronary Stent System (NECSS) was able to be delivered to the target lesion in 100% of cases.
Arm/Group | Acute Success
Number analyzed (Participants) | 49
Participants | 49

2. Secondary Outcome: Physician Assessment Was Performed After Each Case
Description: A short questionnaire about device performance was included in the CRF. Device performance characteristics were rated on a scale of 1 to 5 (1 being poor performance and 5 being excellent performance).
Time Frame: Post procedure
Population: Device preparation
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Patient Receiving the DESyne X2 Coronary Stent: Physician reported scoring system using a rating scale of 1-5 was used, with 1 as poor and 5 as excellent
Arm/Group | Patient Receiving the DESyne X2 Coronary Stent
Number analyzed (Participants) | 49
score on a scale
  Device Preparation | 4.6 [4 to 5]
  Stent System Movement through Guiding Catheter | 4.6 [3 to 5]
  System track and flexibility | 4.3 [3 to 5]
  Stent Positioning | 4.4 [3 to 5]
  Stent and system visibility under Fluoroscopy/cine | 4.5 [4 to 5]
  Delivery system deployment of stent | 4.4 [4 to 5]
  Stent expansion to desired diameter | 4.3 [3 to 5]
  Stent recoil | 4.4 [2 to 5]
  Stent conformability to vessel curvature | 4.3 [3 to 5]
  Delivery system withdrawal through stent and guide catheter | 4.5 [4 to 5]
  Stent re-cross of post dilatation catheter (as appropriate) | 4.3 [4 to 5]

ADVERSE EVENTS:
Time Frame: Peri-procedurally
Groups:
- Patients Receiving the DESyne X2 Coronary Stent: There were 3 reported procedure complications including 2 cases of edge dissection treated with an additional DESyne X2 stent, and 1 case of a guidewire perforation in a non-target vessel during a non-target lesion treatment.
Arm/Group | Patients Receiving the DESyne X2 Coronary Stent
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 3/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Receiving the DESyne X2 Coronary Stent (N=49)
procedure complication (Cardiac disorders) | 2 (2) — edge dissection requiring additional stent placement
guidewire perforation (Cardiac disorders) | 1 (1) — guidewire perforation in a non-target vessel

LIMITATIONS AND CAVEATS:
The study was halted early with enrollment of 49 of the planned 100 patients due to slow enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/85/NCT04375085/Prot_SAP_ICF_001.pdf